CLINICAL TRIAL: NCT01572090
Title: Comparison of Weight Loss Induced by Bariatric Surgery vs Conventional Treatment on Body Composition, Adipokines, Gastro-intestinal Hormones and Cardiometabolic Risk Factors
Brief Title: Comparison of Weight Loss Induced by Bariatric Surgery vs Conventional Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Gema Frühbeck Martínez, MD, PhD, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OBECUN-WL-01
Record Dates: First submitted 2012-03-28; First posted 2012-04-05 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
Keywords: Body mass index; Body fat; Obesity; Bariatric surgery; Conventional dietary treatment; Diabetes Mellitus, Type 2; Cardiometabolic risk factors; Inflammation; Adipokines; Gastrointestinal hormones; Comorbidity improvement; Energy intake; Energy expenditure; Physical activity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Inflammation; Motor Activity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Conventional weight loss: CONV-NG (Active Comparator): Obese normoglycemic (NG) patients evidenced by a body fat ≥ 35% in women and ≥ 25% in men and a 2-h oral glucose tolerance test.
  Conventional weight loss will be achieved by "Lifestyle changes" including advice on increasing physical activity and prescription of a hypocaloric diet providing a daily energy deficit of 500-1000 kcal/d as calculated from the determination of the resting energy expenditure through indirect calorimetry (Vmax29, SensorMedics Corporation, Yorba Linda, CA) and multiplication by the physical activity level factor to obtain the individual's total energy expenditure. Regular visits with the dietitian will be scheduled as in the surgical groups.
  Interventions: Behavioral: Lifestyle Changes
- Conventional weight loss: CONV-T2D (Active Comparator): Obese type 2 diabetic (T2D) patients evidenced by a body fat >35% in women and ≥ 25% in men and proven documentation of T2D diagnosis, history and treatment in accordance with good clinical practice.
  Conventional weight loss will be achieved by "Lifestyle changes" including advice on increasing physical activity and prescription of a hypocaloric diet providing a daily energy deficit of 500-1000 kcal/d as calculated from the determination of the resting energy expenditure through indirect calorimetry (Vmax29, SensorMedics Corporation, Yorba Linda, CA) and multiplication by the physical activity level factor to obtain the individual's total energy expenditure. Regular visits with the dietitian will be scheduled as in the surgical groups.
  Interventions: Behavioral: Lifestyle Changes; Other: Adjustment of oral antidiabetics/insulin therapy
- Laparoscopic Sleeve gastrectomy: SG-NG (Active Comparator): The intervention in this arm comprises obese (BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities) normoglycemic (NG) patients (evidenced by a 2-h OGTT) undergoing a sleeve gastrectomy (SG). The Sleeve gastrectomy SG-NG involves the removal of the mayor curvature of the stomach. Via a laparoscopic approach. In addition to the surgery, patients will have regular follow-up with a dietitian and endocrinologist for appropriate counselling on lifestyle changes (diet, physical activity and vitamin/mineral supplementation counselling) following bariatric surgery.
  Interventions: Behavioral: Lifestyle Changes; Procedure: Laparoscopic sleeve gastrectomy
- Laparoscopic Sleeve gastrectomy: SG-T2D (Active Comparator): The intervention in this arm comprises obese (BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities) type 2 diabetic (T2D) patients with proven documentation of T2D diagnosis, history and treatment in accordance with good clinical practice undergoing a sleeve gastrectomy (SG). In addition to the surgery, patients will have regular follow-up with a dietitian and endocrinologist for appropriate counselling on lifestyle changes (diet, physical activity and vitamin/mineral supplementation counselling) following bariatric surgery as well for adjustment of antidiabetic medication. Adjustment of oral antidiabetics/insulin therapy consisting in continuation, adjustment or discontinuation of medical antidiabetic therapy if needed in accordance with good clinical practice.
  Interventions: Behavioral: Lifestyle Changes; Other: Adjustment of oral antidiabetics/insulin therapy; Procedure: Laparoscopic sleeve gastrectomy
- Laparoscopic R-Y gastric bypass: RYGB-NG (Active Comparator): The intervention in this arm comprises obese (BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities) normoglycemic (NG) patients (evidenced by a 2-h OGTT) undergoing laparoscopic Roux-en-Y gastric bypass (RYGB). In addition to the surgery, patients will have regular follow-up with a dietitian and endocrinologist for appropriate counselling on lifestyle changes (diet, physical activity and vitamin/mineral supplementation counselling) following bariatric surgery.
  Interventions: Behavioral: Lifestyle Changes; Procedure: Laparoscopic Roux-en-Y gastric bypass
- Laparoscopic R-Y gastric bypss: RYGB-T2D (Active Comparator): The intervention in this arm comprises obese (BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities) type 2 diabetic (T2D) patients with proven documentation of T2D diagnosis, history and treatment in accordance with good clinical practice undergoing laparoscopic Roux-en-Y gastric bypass (RYGB). In addition to the surgery, patients will have regular follow-up with a dietitian and endocrinologist for appropriate counselling on lifestyle changes (diet, physical activity and vitamin/mineral supplementation counselling) following bariatric surgery as well for adjustment of antidiabetic medication. Adjustment of oral antidiabetics/insulin therapy consisting in continuation, adjustment or discontinuation of medical antidiabetic therapy if needed in accordance with good clinical practice.
  Interventions: Behavioral: Lifestyle Changes; Other: Adjustment of oral antidiabetics/insulin therapy; Procedure: Laparoscopic Roux-en-Y gastric bypass

INTERVENTIONS:
Behavioral: Lifestyle Changes — Hypocaloric diet providing a 1000 kcal/d deficit from total energy expenditure assessed by indirect calorimetry and physical activity determination.
  Dietetic and physical activity counselling with a dietitian.
  Other Names: Conventional weight loss
Other: Adjustment of oral antidiabetics/insulin therapy — Continuation-discontinuation of medical antidiabetic therapy if needed in accordance with good clinical practice. In addition to the surgery, patients will have regular follow-up with an endocrinologist for appropriate counselling on lifestyle changes (diet, physical activity and vitamin/mineral supplementation counselling) following bariatric surgery as well for adjustment of antidiabetic medication. Adjustment of oral antidiabetics/insulin therapy consisting in continuation, adjustment or discontinuation of medical antidiabetic therapy if needed in accordance with good clinical practice.
  Other Names: Pharmacological treatment adjustment
  Arms: Conventional weight loss: CONV-T2D; Laparoscopic R-Y gastric bypss: RYGB-T2D; Laparoscopic Sleeve gastrectomy: SG-T2D
Procedure: Laparoscopic sleeve gastrectomy — The Laparoscopic sleeve gastrectomy SG-NG involves the removal of the mayor curvature of the stomach via a laparoscopic approach. In addition to the surgery, patients will have regular follow-up with a dietitian and endocrinologist for appropriate counselling on lifestyle changes (diet, physical activity and vitamin/mineral supplementation counselling) following bariatric surgery.
  Other Names: Restrictive bariatric surgery; Laparoscopic sleeve gastrectomy SG
  Arms: Laparoscopic Sleeve gastrectomy: SG-NG; Laparoscopic Sleeve gastrectomy: SG-T2D
Procedure: Laparoscopic Roux-en-Y gastric bypass — Laparoscopic Roux-en-Y gastric bypass. In addition to the surgery, patients will have regular follow-up with a dietitian and endocrinologist for appropriate counselling on lifestyle changes (diet, physical activity and vitamin/mineral supplementation counselling) following bariatric surgery.
  Other Names: Mixed (restrictive & malabsorptive) bariatric surgery
  Arms: Laparoscopic R-Y gastric bypass: RYGB-NG; Laparoscopic R-Y gastric bypss: RYGB-T2D

SUMMARY:
Patients with overweight or obesity are in need to loose weight and represent a particularly challenging medical condition. Undoubtedly, any intervention achieving a negative energy balance over an extended time period will result in weight loss. Although several treatment modalities are available, currently the most extended approaches are lifestyle changes, pharmacotherapy, and bariatric surgery. Given the limited approved anti-obesity drugs, the main therapeutic strategies involve either conventional treatment or bariatric surgery. Conventional weight-reduction programs pursue a safe weight loss rate of 0,5-1,0 kg per week. The main modifiable factors affecting energy balance are dietary energy intake and energy expended through physical activity. In spite of the difficulty in achieving relevant and sustained weight loss via the conventional approach, some patients are successful in reducing weight and obesity-associated complications. Bariatric surgery has proved to be the most effective long-term treatment for weight loss and comorbidity improvement. While some of the surgery-induced benefits are directly dependent on adipose tissue reduction, others are due to specific gastrointestinal changes that take place early on and before any significant effects on body weight are observed. The present study contemplates the determination and comparison of the anthropometric and metabolic changes produced by the conventional and surgery-induced treatment modalities. Particular emphasis will be placed on the potential differential effects between conventional and surgical weight loss on body composition changes, circulating adipokines and gastrointestinal hormones together with their subsequent impact on cardiometabolic risk factors.

DETAILED DESCRIPTION:
In spite of the recognition of obesity as a serious public health problem due to its well-known increased risk for the development of type 2 diabetes hypertension, coronary heart disease, sleep-breathing disorders, and certain forms of cancer, among others, it is proving extraordinarily difficult to halt this pandemia. Strictly speaking obesity does not refer to an excess weight or weight to height ratio. In fact, the World Health Organization defines obesity as a state of increased adipose tissue of sufficient magnitude to produce adverse health consequences. Thus, in order to better define the effects and benefits of weight loss it is important to address the impact on body fat changes. Given the limited approved anti-obesity drugs, the main therapeutic strategies involve either conventional treatment or bariatric surgery. The main modifiable factors affecting energy balance are dietary energy intake and energy expended through physical activity. In spite of the difficulty in achieving relevant and sustained weight loss via the conventional approach, some patients are successful in reducing weight and obesity-associated complications. Bariatric surgery has proved to be the most effective long-term treatment for weight loss and comorbidity improvement. While some of the surgery-induced benefits are directly dependent on adipose tissue reduction, others are due to specific gastrointestinal changes that take place early on and before any significant effects on body weight are observed. Noteworthy, currently available bariatric procedures differ on their impact on these aspects. The present study contemplates the determination and comparison of the anthropometric and metabolic changes produced by the conventional and surgery-induced treatment modalities. Particular emphasis will be placed on the potential differential effects between conventional and surgical weight loss on energy intake, energy expenditure, body composition changes, circulating adipokines and gastrointestinal hormones together with their subsequent impact on cardiometabolic risk factors. The conventional weight-reduction program (CONV) will pursue a safe weight loss rate of 0,5-1,0 kg per week. The surgery-induced weight loss will be achieved by two of the most frequently used bariatric operations, the sleeve gastrectomy [SG (which implies a restrictive component)] and the Roux-en-Y gastric bypass [RYGB (which combines a restrictive and a malabsorptive component)].

The purpose of the study is to determine the effect of three weight loss procedures that differ on their manipulation of the anatomical and functional characteristics of the gastrointestinal tract. While in the conventional treatment the gastrointestinal system remains intact, in the SG only the stomach is manipulated as opposed to the RYGB, where both the stomach and the small intestine are operated on. Since bariatric surgery is well known to induce partial or total remission of type 2 diabetes mellitus, the effects of the three different weight loss procedures will be assessed separately in obese normoglycemic and obese type 2 diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65 years.
* Obesity as defined by World Health Organization criteria.
* For bariatric surgery patients: qualified for obesity surgery by the -Multidisciplinary Obesity Team of the Clinica Universidad de Navarra
* For type 2 diabetic patients: T2D diagnosis confirmed by either fasting plasma glucose ≥126 mg/dL on two separate occasions, or fasting plasma glucose ≥126 mg/dL and plasma glucose ≥140 mg/dL 2 h after OGTT, or treatment with anti-diabetic medication in accordance with good clinical practice with and well-documented information on diagnosis, history, treatment(s) and HbA1c data.
* No major organ disease unrelated to excess body weight.
* Mentally able to understand the study and willingness to participate in the study.

Exclusion Criteria:

* Pregnancy/lactation
* Poor overall general health
* Drug and/or alcohol addiction
* Prior bariatric or gastrointestinal surgery
* Active gastric or intestinal tract disease
* Thyroid disease
* Type 1 diabetes mellitus
* Portal hypertension and/or cirrhosis
* Malignancies
* History of eating disorders or major psychiatric illness
* Unable to communicate with study staff

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in body fat | Baseline, 1, 6, 12, and 24 months
  Body fat will be assessed by air-displacement plethysmography (Bod-Pod) over the duration of the intervention.

SECONDARY OUTCOMES:
Change in energy balance | Baseline, 1, 6, 12 and 24 months
  Energy intake will be assessed by food dietary, 24-h recall, FFQ and energy expenditure will be determined by indirect calorimetry, physical activity questionnaires and accelerometry over the duration of the intervention.
Change in glycemic control | Baseline, 1, 6, 12 and 24 months
  Measurement of fasting plasma glucose, insulin and HbA1c concentrations over the duration of the intervention.
Change in cardiovascular risk factors | Baseline, 1, 6, 12 and 24 months
  Measurement of circulating total cholesterol, LDL-cholesterol, HDL-cholesterol, fibrinogen, C-reactive protein, homocysteine, von Willebrand factor and adipokines over the duration of the intervention.
Change in gastrointestinal hormones | Baseline, 1, 6, 12 and 24 months
  Measurement of fasting ghrelin, PYY, GLP-1, GIP, PP, amylin and oxyntomodulin over the duration of the intervention.
Change in gustatory threshold | Baseline, 1, 6, 12 and 24 months
  Determination of the gustatory threshold levels by the whole-mouth chemical test procedure and tongue electrogustometry over the duration of the intervention.
Change in BMI | Baseline, 1, 6, 12 and 24 months
  Measurement of weight and height over the duration of the intervention to calculate the BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Gema Frühbeck, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez-Ambrosi J, Gonzalez-Crespo I, Catalan V, Rodriguez A, Moncada R, Valenti V, Romero S, Ramirez B, Silva C, Gil MJ, Salvador J, Benito A, Colina I, Fruhbeck G. Clinical usefulness of abdominal bioimpedance (ViScan) in the determination of visceral fat and its application in the diagnosis and management of obesity and its comorbidities. Clin Nutr. 2018 Apr;37(2):580-589. doi: 10.1016/j.clnu.2017.01.010. Epub 2017 Jan 28. PMID 28187933
- [Derived] Gomez-Ambrosi J, Gallego-Escuredo JM, Catalan V, Rodriguez A, Domingo P, Moncada R, Valenti V, Salvador J, Giralt M, Villarroya F, Fruhbeck G. FGF19 and FGF21 serum concentrations in human obesity and type 2 diabetes behave differently after diet- or surgically-induced weight loss. Clin Nutr. 2017 Jun;36(3):861-868. doi: 10.1016/j.clnu.2016.04.027. Epub 2016 May 4. PMID 27188262